CLINICAL TRIAL: NCT01905878
Title: Biological Half Life of DLBS1033 in Healthy Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: Dexa Medica Group (Industry)
Responsible Party: Principal Investigator, Melva Louisa, SSi, M. Biomed, Doctor, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: halflifeDLBS1033
Record Dates: First submitted 2013-07-11; First posted 2013-07-23 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Healthy Condition
MeSH Terms: interventions — DLBS 1033

STUDY DESIGN:
Intervention Model Description: This study was open label-single arm trial, which was done at Pharmacology and Therapeutic Department and Clinical Pathologic Department of Faculty Medicine of University of Indonesia Cipto Mangunkusumo Hospital. The study drug was enteric coated DLBS1033 tablet, which contained 490 mg bioactive protein fraction; and produced by PT Dexa Medica, Tangerang, Indonesia.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- single dose DLBS1033 (Experimental): Before taking the drug, blood samples will be collected from subject to assess PAP complex level, serum creatinine, SGOT, SGPT, PT and aPTT. After that, subjects will instructed to take three tablets enteric coated of DLBS1033 in front of investigator. After take the medicine blood sample will be collected on 30 minute, 60 minute, 90 minute, 2 hour, 3 hour, 4 hour, 6 hour, 8 hour, 10 hour, 12 hour, and 24 hour to evaluate serial PAP complex. Subjects will undergo a clinical assessment including vital signs and the presence of adverse events at the time of blood sampling. On this trial, subjects are only permitted to eat food from investigator.
  Interventions: Drug: DLBS1033
- steady state of DLBS1033 (Experimental): On day 1 blood samples will be collected to assess PAP complex level, serum creatinine, SGOT, SGPT, PT and aPTT. After that, subjects will instructed to take one tablet of DLBS1033 in front of investigator. Study drug packages (that consist of 8 tablets) will dispense to the subjects at day-1 and instructed to take the drug 3 times daily 30 minutes before meals. Subjects also will instructed to record any adverse events and concomitant medication prescribed in diary card. Subjects have to take the drug on 3 days (day 1, 2, and 3). On day 4, blood sample will be collected on 0 minutes, 30 minute, 60 minute, 90 minute, 2 hour, 3 hour, 4 hour, 6 hour, 8 hour, 10 hour, 12 hour, and 24 hour to evaluate serial PAP complex. Subjects will undergo a clinical assessment including vital signs and the presence of adverse events at the time of blood sampling. On this trial, subjects are only permitted to eat food from investigator.
  Interventions: Drug: DLBS1033

INTERVENTIONS:
Drug: DLBS1033

SUMMARY:
DLBS1033 is bioactive protein fraction which extracted from Lumbricus rubellus earthworm. This earthworm comes from Pengalengan, West Java, Indonesia. DLBS1033 possesses 8 major proteins with molecular weight below 100 kDa, so its named as Lumbricus Low Molecular weight Proteins (LLP). This enzyme can be transported to the bloodstream via intestinal epitel. As a drug that consists of serin protease enzyme, suspected that the mechanism of action of lumbrokinase, especially as fibrinolytic and antithrombotic. One study of DLBS1033 concluded that plasmin-antiplasmin (PAP) complex is a sensitive parameter for evaluating fibrinolytic effect of this drug. But, until now there is no clinical study that evaluate pharmacokinetic of this drug. As a pilot study, the aim of this study is to evaluate biological half life of DLBS1033.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18-55 years old
* Body mass index between 18-25 kg/m2
* Normal physical examination
* Patient still have the ability to undergo examinations and give written informed consent
* Plasmin-antiplasmin complex (PAP complex) level between 0-514 ng/ml

Exclusion Criteria:

* Patient with cardiovascular disease, hypertension, diabetes mellitus, and dyslipidemia
* Creatinin serum more than 1,5 x ULN
* SGOT and SGPT more than 3 x ULN
* Blood pressure ≥ 140/90 mmHg
* Fasting blood glucose > 126 mg/dL
* Alcohol patients
* Took any medications (including traditional medicine, supplement and vitamin) in 1 week before the study)
* Patient has bleeding history which unclear etiology
* Hemoglobin < 10 g/dL
* Thrombocyte count < 100.000/microliter
* Heavy smoker (Bringman Index > 600)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Serial Plasmin-antiplasmin complex (PAP complex) | 3 days
  PAP complex will be measured on 0 minute, 30 minute, 60 minute, 90 minute, 2 hour, 3 hour, 4 hour, 6 hour, 8 hour, 10 hour, 12 hour, and 24 hour

CONTACTS AND LOCATIONS:
Overall Officials: Anggi Gayatri, MD, SpFK, Principal Investigator — Indonesia University
Locations (1):
- University of Indonesia, Jakarta, Indonesia